CLINICAL TRIAL: NCT02756780
Title: Tenovus Cancer Choirs: the Effect of Choir Singing on Psychological and Immune Responses of Cancer Patients, Staff and Carers
Brief Title: Tenovus Cancer Choirs Study: the Benefits of Singing for Those Affected by Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: London Cancer Alliance (Unknown); Royal College of Music (Other); Tenovus Cancer Care (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SWU2016
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: Remission; Carer; Psychological; Bereaved; Cancer; Breast; Prostate; Colorectal; Music
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenovus Cancer Choir (Experimental): Participants will be asked to attend 12 weeks of weekly choir rehearsals lasting approximately 1 hour. Following the first 12 weeks, participants will no longer be asked to attend rehearsals, but are welcome to do so. Whether or not they do and how many they attend will be measured as an outcome variable to assess whether initial 3-month involvement leads to long-term engagement.
  Interventions: Other: Tenovus Cancer Choir
- Control (no choir) Group (No Intervention): If eligible participants are unable to make the dates and times or live too far away but fulfil all the same criteria (including expressing an interest in singing) they will become part of the control group. This will involve the same data collection as the Cancer Choir Group but participants will not sing in a weekly choir.

INTERVENTIONS:
Other: Tenovus Cancer Choir — Choir sessions will take place at both of the Royal Marsden Hospital sites on a weekly basis. Sessions typically consist of learning popular songs with messages of support. Songs are learnt without sheet music, using specially created backing tracks. These are also made available to participants at home so they can continue singing away from the sessions. No singing experience is required and the main aim of the sessions is enjoyment and meeting other people. Sessions will take place in the early evening so that participants have the option of staying to socialise afterwards.
  Arms: Tenovus Cancer Choir

SUMMARY:
'Sing With Us' choirs are an initiative established in Wales by Tenovus Cancer Care to provide social support and improve mental wellbeing amongst those affected by cancer, whether patients, carers or staff. Research has already demonstrated that these choirs can reduce depression and anxiety amongst participants and improve social support networks and quality of life as well as preliminary evidence that they can reduce levels of stress hormones and improve immune function. The aim of this study is to establish more about the psychological benefits of regular choir singing and explore whether the biological changes noted in pilot studies can be sustained over time. This could identify whether choirs have the potential to optimise health in people affected by cancer, helping to put patients in the best position to receive treatment or maintain remission and supporting those who care for someone with cancer, whether professionally or informally.

DETAILED DESCRIPTION:
There is growing evidence that psychosocial interventions from mindfulness to yoga to the arts can reduce symptoms of depression and anxiety, increase social support networks, improve quality of life and raise perceptions of care in people affected by cancer 1,2. These positive states have, in turn, been linked with optimised immune responses including reduced stress hormones and enhanced cellular activity 1,3,4. However, despite growing numbers of music interventions for cancer care, there is little research into their psychobiological impact.

'Sing With Us' choirs are an initiative established in Wales by Tenovus Cancer Care to provide social support and improve mental wellbeing amongst those affected by cancer, whether patients, carers or staff. Research has already demonstrated that these choirs can reduce depression and anxiety amongst participants and improve social support networks and quality of life as well as preliminary evidence that they can reduce levels of stress hormones and enhance immune activity 5,6. The aim of this study is to establish more about the psychological benefits of regular choir singing and explore whether the biological changes noted in pilot studies can be sustained over time. This could identify whether choirs have the potential to optimise health in people affected by cancer, helping to put patients in the best position to receive treatment or maintain re mission and supporting those who care for someone with cancer, whether professionally or informally.

As part of this project, and in addition to the choirs already run by Tenovus Cancer Care, Tenovus will fund two choirs, one at each of the Royal Marsden sites. These will run on a weekly basis for 18 months and will consist of a session lasting 1 hour led by a professional choir leader who is a member of the Tenovus Cancer Care staff. The choirs will be open to anybody affected by cancer at the Royal Marsden Hospital or in the local area. However, there will be three cohorts of patients involved in the research running alongside the choir: cohorts A and B involving active recruitment of participants and Cohort C in which people who join the choir of their own volition but are not eligible for the first 3 cohorts will be invited to participate:

Cohort A: breast, prostate and colorectal cancer patients will be invited to join the study for a period of 12 weeks. If they are able to make the dates and times of the choir sessions they will become part of the experimental group. If they are unable to make the dates and times or live too far away but fulfil all the same criteria (including expressing an interest in singing) they will become part of the control group. Data collection for all participants will include (a) completing psychological scales which will be available in hard copy or as online versions; (b) providing saliva samples before 4 choir rehearsals: week 1, week 6 and week 12 with a three month follow-up (week 24). Experimental participants will be expected to attend as many of the first 12 choir sessions in the time period as possible but will then select whether they continue involvement in the choir for the following 12 weeks.

Cohort B: hospital staff, carers of somebody affected by cancer and bereaved carers will be invited to join the study for a period of 12 weeks. Recruitment and participation for this Cohort (including the presence of a control group) will be as in Cohort A except there will be no biological component. Participants will merely complete the online psychological questionnaires.

Cohort C: all other participants who decide to join the choirs (whether patients, carers or staff) will be invited to take part in the psychological part of the study, completing the anonymous questionnaires at weeks 0, 6, 12 and 24. This will be an uncontrolled Cohort. But it may identify additional participant groups for whom the choirs provide support.

ELIGIBILITY:
Inclusion Criteria:

* COHORT A: (i) Patients with stage I-III breast cancer up to 24 months post diagnosis
* (ii) Patients with diagnosed prostate cancer on active surveillance
* (iii) Patients with colorectal cancer stages I-III up to 24 months post diagnosis
* COHORT B: (i) Members of staff at a hospital
* (ii) People who care for somebody with cancer, whether formally or informally
* (iii) People who have lost a family member or somebody they cared for to cancer in the last 3 years
* COHORT C: anybody who is affected by cancer and has joined the choir

General exclusion Criteria:

* Participants aged under the age of 18
* Level of English insufficient to provide informed consent or complete the psychological questionnaires
* Refusal to participate
* Already engaged in a weekly group choir
* Started a formal course of psychological therapy in the past 1 month or scheduled to start in the next 12 weeks
* Started any new medication for anxiety or depression in the last month

Additional exclusion criteria for cohort A:

* Currently having chemotherapy or radiotherapy or less than 90 days since last session
* Scheduled for surgery in the next 12 weeks or less than 90 days post surgery
* Have a current diagnosis of an additional immune condition e.g. lupus
* Currently being treated with steroids or immunosuppressive medication
* Participants who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Anxiety & Depression | Change in anxiety and depression level at weeks 6, 12 and 24 compared to baseline
  Hospital Anxiety and Depression Scale (HADS)

SECONDARY OUTCOMES:
Social Support | Change in social provision level at weeks 6, 12 and 24 compared to baseline
  Social Provisions Scale (SPS)
Wellbeing | Change in wellbeing level at weeks 6, 12 and 24 compared to baseline
  Warwick-Edinburgh Short Questionnaire (WEMWBS)
Self-efficacy | Change in self-efficacy level at weeks 6, 12 and 24 compared to baseline
  General Self-Efficacy scale short form (GSE-6)
Self-esteem | Change in self-esteem level at weeks 6, 12 and 24 compared to baseline
  Sing Item Self-Esteem Scale
General Health | Change in general health level at weeks 6, 12 and 24 compared to baseline
  Short Form 12 Health Survey (SF12)
Stress hormones | Change in stress hormone levels at weeks 6, 12 and 24 compared to baseline
  Salivary cortisol levels
Immune proteins | Change in immune protein levels at weeks 6, 12 and 24 compared to baseline
  Saliva cytokines, chemokines and receptors

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Wiseman, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London/Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fancourt D, Finn S, Warran K, Wiseman T. Group singing in bereavement: effects on mental health, self-efficacy, self-esteem and well-being. BMJ Support Palliat Care. 2022 Oct;12(e4):e607-e615. doi: 10.1136/bmjspcare-2018-001642. Epub 2019 Jun 26. PMID 31243022